CLINICAL TRIAL: NCT01688401
Title: Intra-arterial Chemotherapy for the Treatment of Progressive Diffuse Intrinsic Pontine Gliomas (DIPG).
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Solving Kids' Cancer (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: J11164; NA_00069122 (Other: JHMIRB)
Record Dates: First submitted 2012-09-10; First posted 2012-09-19 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Diffuse Intrinsic Pontine Glioma (DIPG)
Keywords: diffuse intrinsic pontine glioma (DIPG); intra-arterial chemotherapy; angiography
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma | interventions — Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IA melphalan (Experimental): IA melphalan is administered via the basilar artery.
  Interventions: Drug: Melphalan hydrochloride

INTERVENTIONS:
Drug: Melphalan hydrochloride — Drug administered intra-arterially (injection in the artery).
  Standard dose: Cycle 1: 1 mg, intra-arterial (IA) delivery. Cycle 2: 2 mg, intra-arterial (IA) delivery.
  Duration of treatment: Eight weeks total - two cycles of IA chemotherapy, separated by four weeks.
  Other Names: Alkeran

SUMMARY:
The goal of this pilot study is to determine if intra-arterial (IA) chemotherapy is safe in the treatment of progressive diffuse intrinsic pontine gliomas (DIPG). IA administration of the chemotherapeutic agent enhances the regional distribution of the drug, thereby increasing the local delivered dose while minimizing systemic toxicity. It also provides a treatment option for these patients at the time of tumor recurrence.

DETAILED DESCRIPTION:
Delivering the chemotherapeutic agent directly to the tumor via the arterial system avoids the complications and adverse events associated with toxicity from systemic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients of all ages with progressive DIPG.
* Consensus following presentation of the case at the multidisciplinary Pediatric Neuro-Oncology conference, which includes participation of neuro-oncology, neurosurgery, radiation oncology, interventional neuroradiology and neurology.

Exclusion Criteria:

* Documented hypercoagulable disorders or vasculopathies

  * INR value more than a Grade 1 toxicity by CTCAE v 4.0 criteria (>1 - 1.5 x ULN; >1 - 1.5 times above baseline if on anticoagulation).
  * APTT value more than a Grade 1 toxicity by CTCAE v 4.0 criteria (>ULN - 1.5 x ULN).
* Platelets less than 50 x 103/mm3
* Absolute neutrophil count less than 500/ mm3
* Pregnancy
* Documented severe allergic reaction to IV iodinated contrast, specifically bronchospasm and anaphylaxis.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2013-03-08 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2018-11-26 (Actual)

PRIMARY OUTCOMES:
Technical safety as determined by number of participants with toxicity | 60 days
  Number of participants with grades 3-5 intracranial hemorrhage, grades 3-5 stroke, as defined by the Nervous system disorder CTCAE, and requirement of blood transfusion.

SECONDARY OUTCOMES:
Long-term Efficacy as assessed by progression free survival | 2 years
  Number of months until disease progression.

OTHER OUTCOMES:
Immediate Efficacy as assessed by number of participants with decrease in required steroid dose | 60 days
Immediate Efficacy as assessed by number of participants with decrease in tumor size on MRI | 60 days
Immediate Efficacy as assessed by number of participants with decrease in the degree of enhancement on MRI | 60 days
Immediate Efficacy as assessed by number of participants with improved neurological examination | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Monica Pearl, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States